CLINICAL TRIAL: NCT05332587
Title: Efficacy and Safety of Low-dose Rituximab in the Treatment of Refractory Myasthenia Gravis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu Weibin, Director of Neurology Department, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2020]414-1
Record Dates: First submitted 2021-12-04; First posted 2022-04-18 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Refractory Myasthenia Gravis; Rituximab
MeSH Terms: conditions — Myasthenia Gravis | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab Treated (Experimental): rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — The therapeutical schema is rituximab 100-200 mg/week for a total of 2-4 times

SUMMARY:
This study is designed to evaluate the effectiveness and safety of low-dose rituximab in patients with refractory myasthenia gravis.

The traditional treatment of MG is immunosuppressive therapy, usually beginning with corticosteroids. However, up to 70% of treated patients show an incomplete response, including 10 - 30% who are unresponsive. Corticosteroids and other immunosuppressive therapies presented also many side effects. The investigators propose to evaluate in a pilot, open, prospective, single central study, the interest of rituximab (RTX) in the treatment of patients with refractory MG. Fifty patients with refractory MG will be included in the study and divided into two stages: 14 patients in the first stage were followed up after using RTX according to the study protocol. The study will move into the second stage on if the number of effective cases is greater than 3, otherwise, the study will be discontinued (based on Simon's Optimal Two-stage Design). The remaining 36 patients were enrolled in the second stage. In the first and second stages, the treatment plan and follow-up plan were consistent. The therapeutical schema is rituximab 100-200 mg/week for a total of 2-4 times, followed by adequate organ function, laboratory parameters and assessment of MG after each injection and end of follow up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 80 and under;
2. Myasthenia gravis:

   1. Patients who are diagnosed as generalized or ocular myasthenia gravis
   2. Patients must have disease refractory to treatment: the condition did not improve (QMG score decreased by less than 3 points after treatment) or even deteriorated after treatment with sufficient prednisone or other immunosuppressive agents.
3. Patients sign informed consent forms

Exclusion Criteria:

1. Over the age of 80
2. Patients with serious complications such as infection
3. Patients with active TB (during the screening period, a chest X-ray or chest CT would be performed unless the patient can provide chest X-ray or chest CT reports in the last month); or patients with active HBV, HBV DNA> 200
4. Patients suffering from cardiomyopathy, acute coronary events, or severe arrhythmia.
5. Patients who were allergic to rituximab
6. Pregnant or suckling period woman
7. Patients accompanied with mental disorders and have difficult to communication
8. Patients with a significant abnormality in white blood cells, hemoglobin, and platelet count.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to reach MM-1, the proportion of drug remission. | 27 weeks
  Mild clinical Manifestations（MM-1）was the primary efficacy endpoint observed. Record the time the patient appears from the time of medication to the time of MM-1，and calculate the percentage of Pharmacologic Remission (PR). Criteria for PR: The patient has had no symptoms or signs of MG and continues to take some form of therapy for MG. There is no weakness of any muscle on careful examination by someone skilled in the evaluation of neuromuscular disease. Isolated weakness of eyelid closure is accepted. Patients taking cholinesterase inhibitors are excluded from this category because their use suggests the presence of weakness.

SECONDARY OUTCOMES:
The changes of the disease severity | 27 weeks
  The magnitude by which the Quantitative Myasthenia Gravis (QMG) (0-39), the Myasthenia Gravis-specific Activities of Daily Living scale (MG-ADL) (0-24) , the MG Composite (MGC) (0-46) or the MG 15-item Quality of Life scale (MG-QOL15) (0-60) scores are changed. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, China